CLINICAL TRIAL: NCT05624138
Title: The Possible Protective Role of Ketotifen Against Oxaliplatin Induced Peripheral Neuropathy in Patients With Colorectal Cancer
Brief Title: The Possible Protective Role of Ketotifen Against Oxaliplatin Induced Peripheral Neuropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Salma Samah Sayed Wahby, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ketotifen in neuropathy
Record Dates: First submitted 2022-11-08; First posted 2022-11-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Ketotifen

STUDY DESIGN:
Intervention Model Description: - Study design This study will be a Randomized placebo controlled parallel study Group one (Placebo group or code A; n=32)
  Patients will receive 12 cycles of modified FOLFOX-6 regiment plus placebo tablets daily throughout the twelve chemotherapy cycles. The chemotherapy cycles will be received every 2 weeks and will be as follows:
  Day 1: Oxaliplatin 85 mg/m2 intravenous infusion in 250-500 mL 5% dextrose solution and leucovorin 400 mg/m2 intravenous infusion in 5% dextrose solution both were given over 120 minutes at the same time in separate bags using a Y-line access, followed by 5-fluorouracil 400 mg/m2 intravenous bolus given over 2-4 minutes, followed by 5-fluorouracil 2400 mg/m2 intravenous infusion in 500 mL 5% dextrose solution as a 46-hour infusion.
  Group two (Ketotifen group or code B; n=32) Patients will receive the same chemotherapy regimen as group one in addition to oral ketotifen 2 mg daily throughout the twelve chemotherapy cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Group I Placebo group n=32 Patients will receive 12 cycles of modified FOLFOX-6 regiment plus placebo tablets 2mg daily throughout the twelve chemotherapy cycles. The chemotherapy cycles will be received every 2 weeks and will be as follows:
  Day 1 and Day 15: Oxaliplatin 85 mg/m2 intravenous infusion in 250-500 mL 5% dextrose solution and leucovorin 400 mg/m2 intravenous infusion in 5% dextrose solution both were given over 120 minutes at the same time in separate bags using a Y-line access, followed by 5-fluorouracil 400 mg/m2 intravenous bolus given over 2-4 minutes, followed by 5-fluorouracil 2400 mg/m2 intravenous infusion in 500 mL 5% dextrose solution as a 46-hour infusion.
  Interventions: Drug: Placebo tablets
- ketotifen oral tablets (Active Comparator): Group II ketotifen group n=32 Patients will receive 12 cycles of modified FOLFOX-6 regiment plus ketotifen tablets 2mg daily throughout the twelve chemotherapy cycles. The chemotherapy cycles will be received every 2 weeks and will be as follows:
  Day 1 and Day 15 : Oxaliplatin 85 mg/m2 intravenous infusion in 250-500 mL 5% dextrose solution and leucovorin 400 mg/m2 intravenous infusion in 5% dextrose solution both were given over 120 minutes at the same time in separate bags using a Y-line access, followed by 5-fluorouracil 400 mg/m2 intravenous bolus given over 2-4 minutes, followed by 5-fluorouracil 2400 mg/m2 intravenous infusion in 500 mL 5% dextrose solution as a 46-hour infusion
  Interventions: Drug: Ketotifen Oral Tablet

INTERVENTIONS:
Drug: Placebo tablets — 12 cycles of modified FOLFOX-6 regimen (Oxaliplatin, Fluorouracil, calcium leucovorin) with 2 mg placebo tablets
  Other Names: Oxaliplatin, Fluorouracil, calcium leucovorin
  Arms: placebo
Drug: Ketotifen Oral Tablet — ketotifen is a potent anti histaminic drug that may prevent oxaliplatin induced peripheral neuropathy and mucositis and will be administered 2 mg daily along with the 12 cycles of modified Folfox-6 regimen
  Other Names: ketotifen
  Arms: ketotifen oral tablets

SUMMARY:
The aim of current study is to evaluate the possible protective role of Ketotifen against oxaliplatin-induced peripheral sensory neuropathy in patient with stage III colorectal cancer.

This study will be a randomized placebo controlled parallel study.64 patients with colorectal cancer will be randomized to 2 groups:

Group I (control group; n=32) which will receive 12 cycles of modified FOLFOX-6 regimen plus placebo tablets twice daily.

Group II (ketotifen group; n=32) which will receive modified FOLFOX-6 regimen in addition to ketotifen 2 mg daily

Blood sample collection and biochemical assessment:

* Serum IL-6 as a marker of inflammation.
* Serum superoxide dismutase (SOD) as a biomarker of oxidative stress.
* Serum neurotensin as a biomarker for neuropathy.

Assessment of oxaliplatin induced peripheral sensory neuropathy will be done through:

* The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) for grading of neuropathy at baseline and by the end of every two oxaliplatin cycles.
* The use of Neurotoxicity- 12 item questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group "FACT/GOG-Ntx-12" at baseline and by the end of every two oxaliplatin cycles.
* The assessment of the severity of neuropathic pain through brief pain inventory short form "BPI-SF" worst item. Severity of neuropathic pain will be assessed at baseline and by the end of every two oxaliplatin cycles.

DETAILED DESCRIPTION:
The aim of current study is to evaluate the possible protective role of Ketotifen against oxaliplatin-induced peripheral sensory neuropathy in patient with stage III colorectal cancer.

- Study design

This study will be a Randomized placebo controlled parallel study. Sixty four patients with stage III colorectal cancer will be scheduled to receive 12 cycles of modified FOLFOX-6 (folinic acid, flurouracil and oxaliplatin). Patients will be recruited from the Oncology Department, Tanta University Hospital, Tanta, Egypt. Staging will be done according to the American Joint Committee on Cancer 7th edition staging (Edge and Compton, 2010). At admission, patients will be randomized through sealed envelopes method with assignment codes (A and B) into two groups to receive either Placebo or ketotifen in addition to the chemotherapeutic regimen:

Group one (Placebo group or code A; n=32)

Patients will receive 12 cycles of modified FOLFOX-6 regiment plus placebo tablets daily throughout the twelve chemotherapy cycles. The chemotherapy cycles will be received every 2 weeks and will be as follows:

Day 1: Oxaliplatin 85 mg/m2 intravenous infusion in 250-500 mL 5% dextrose solution and leucovorin 400 mg/m2 intravenous infusion in 5% dextrose solution both were given over 120 minutes at the same time in separate bags using a Y-line access, followed by 5-fluorouracil 400 mg/m2 intravenous bolus given over 2-4 minutes, followed by 5-fluorouracil 2400 mg/m2 intravenous infusion in 500 mL 5% dextrose solution as a 46-hour infusion.

Group two (Ketotifen group or code B; n=32) Patients will receive the same chemotherapy regimen as group one in addition to oral ketotifen 2 mg daily throughout the twelve chemotherapy cycles.

Intravenous 5-HT3 antagonist plus pantoprazole will be administered to all participants before each cycle as prophylactic therapy against chemotherapy induced nausea, vomiting and mucositis.

Blood sample collection and biochemical assessment:

* Serum IL-6 as a marker of inflammation.
* Serum superoxide dismutase (SOD) as a biomarker of oxidative stress.
* Serum neurotensin as a biomarker for neuropathy.

Assessment of oxaliplatin induced peripheral sensory neuropathy will be done through:

* The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) for grading of neuropathy at baseline and by the end of every two oxaliplatin cycles.
* The use of Neurotoxicity- 12 item questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group "FACT/GOG-Ntx-12" at baseline and by the end of every two oxaliplatin cycles.
* The assessment of the severity of neuropathic pain through brief pain inventory short form "BPI-SF" worst item. Severity of neuropathic pain will be assessed at baseline and by the end of every two oxaliplatin cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of Stage III colorectal cancer.
* Patients who will be scheduled to receive modified FOLFOX-6.
* Patients with no contraindication to chemotherapy.
* Males and females aged ≥ 18 years old.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate renal function (serum creatinine < 1.5 mg/dl or creatinine clearance (ClCr) ˃ 45 mL/min).
* Patients with adequate liver function (serum bilirubin < 1.5 mg/dl).
* Patients with performance status 0-1 according to Eastern Cooperative Oncology Group (ECOG) score.

Exclusion Criteria:

* Children < 18 years old.
* Prior exposure to neurotoxic chemotherapy (Oxaliplatin, cisplatin, vincristine, paclitaxel, or docetaxel, INH) for at least 6 months prior the study treatment.
* Evidence of pre-existing peripheral neuropathy resulting from another reason (diabetes, brain tumor, brain trauma).
* Patients with diabetes and other conditions that predispose to neuropathy as hypothyroidism, autoimmune diseases, hepatitis C.
* History of known allergy to oxaliplatin or other platinum agents.
* Patients with other inflammatory or stressful conditions.
* Patients with glaucoma, cataract, other chronic eye disease, seizure, diabetes, heart diseases, low blood pressure, dizziness, vertigo, ménière's disease and CNS disorders.
* Concomitant use of multivitamins (vitamins E, C, A), tricyclic antidepressants, other neuro-protective medications (gabapentin, lamotrigine, carbamazepine and phenytoin, etc…).
* Patients on amifampridine, bupropion and donepezil.
* Concurrent active cancer originating from a primary site other than colon or rectum.
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
variation in 12-item neurotoxicity questionnaire (Ntx-12) total score | 6 months (at baseline and after 2 oxaliplatin cycles( the cycle is every 15 days)
  the Ntx-12 questionnaire is comprised of 12 statements intended to measure the severity and impact of peripheral sensory neuropathy on patients' lives. Patients will be instructed to complete the Arabic version of the Ntx-12 and choose the number corresponding to how true each statement was for them using a likert-type scale, with 0 indicating not at all; 1, a little bit; 2, somewhat; 3, quite a bit; and 4, very much
variation in pain rating scale score | 6 months (at baseline and after 2 oxaliplatin cycles( the cycle is every 15 days)
  The assessment of the severity of neuropathic pain through brief pain inventory short form "BPI-SF" worst item. Severity of neuropathic pain will be assessed at baseline and by the end of every two oxaliplatin cycles.
the percentage of patients with peripheral sensory neuropathy grade ≥ 2 | 6 months
  Grading according to National Cancer Institute Common Terminology. there are 5 grades; Grade (1) is asymptomatic may be accompanied by loss of tendon reflex or paresthesia. Grade (2) is moderate symptoms which limit instrumental activities of daily life Grade (3) is severe symptoms which limit self-care activates of daily life. Grade (4) is life threatening consequences or urgent intervention indicated. Grade (5) is death.
  Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017)

SECONDARY OUTCOMES:
changes in serum levels of the measured biological marker Serum IL-6 | 6 months (after 12 cycles and the cycle is every 15 days)
  as a marker of inflammation
changes in serum levels of the measured biological marker Serum SOD | 6 months(after 12 cycles and the cycle is every 15 days)
  as a biomarker of oxidative stress
changes in serum levels of the measured biological marker Serum neurotensin | 6 months ( after 12 cycles and the cycle is every 15 days)
  biomarker for neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology department Tanta university, Tanta, Other, Egypt

IPD SHARING:
Plan to Share IPD: No